CLINICAL TRIAL: NCT06844162
Title: Comparison of Postoperative Analgesic Efficacy of Suprainguinal Fascia Iliaca Block (SFIB) and Pericapsular Nerve Group (PENG) Block With Lateral Femoral Cutaneous Nerve (LFCN) Block in Patients Undergoing Total Hip Arthroplasty
Brief Title: Pericapsular Nerve Group With Lateral Femoral Cutaneous Nerve Block vs Suprainguinal Fascia Iliaca Block for Analgesia in Total Hip Arthroplasty: A Prospective Comparative Study
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güneş Çelebioğlu, Lecturer, Hacettepe University
Other Study IDs: KA-22088
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Coxarthrosis; Primary
Keywords: Suprainguinal fascia iliaca block; PENG block; Lateral femoral cutaneous nerve block; Postoperative analgesia
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SFIB: Patients undergoing THA who received ultrasound-guided SFIB with 0.25% bupivacaine 40 mL under the fascia iliaca with cranial spread.
- PENG: Patients undergoing THA who received ultrasound-guided PENG (0.5% bupivacaine 15 mL) at the iliopubic eminence plus LFCN block (0.5% bupivacaine 5 mL) distal to the inguinal ligament.

SUMMARY:
Prospective observational cohort comparing analgesic efficacy of suprainguinal fascia iliaca block (SFIB) vs pericapsular nerve group block combined with lateral femoral cutaneous nerve block (PENG+LFCN) in primary total hip arthroplasty under general anesthesia (n=48). Outcomes include VAS pain at rest and with movement at 3, 12, 24, 48 h; morphine use (0-3, 3-12, 12-24, 24-48 h; total 0-48 h); quadriceps strength at 6 and 24 h; physiotherapy participation at 24 and 48 h; and adverse events within 48 h.

DETAILED DESCRIPTION:
Adults undergoing primary posterolateral THA under general anesthesia were included if they received either SFIB or PENG+LFCN. Pain (VAS at rest and with 45° passive flexion) was recorded at 3, 12, 24, and 48 h. Morphine via PCA was recorded for 0-3, 3-12, 12-24, and 24-48 h, with a 0-48 h total. Quadriceps strength (0-2 scale) was assessed at 6 and 24 h; physiotherapy participation at 24 and 48 h; opioid- or block-related adverse events through 48 h.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo primary total hip arthroplasty with a diagnosis of coxarthosis

Exclusion Criteria:

* Patients who have a history of neuropathy, patients with renal and hepatic insufficiency, patients with known coagulopathy, patients with a history of allergy to local anesthetics, patients with a history of inguinal surgery on the same side and patients with impaired mental status

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 48 patients of American Society of Anesthesiologists physical status I-II between the age of 18 to 90 years who were scheduled to undergo primary Total hip arthroplasty with a diagnosis of coxarthrosis
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale scores | In the 48 hours following surgery
  Postoperative Visual Analogue Scale scores ( Minimum of 0 and maximum of 10 with higher scores indicative of more severe pain) will be measured at rest and 45 degrees passive flexion at 3, 12, 24 and 48th hours postoperatively

SECONDARY OUTCOMES:
Opioid consumption | In the 48 hours following surgery
  Opioid consumption during 0-3,12-24, 24-48 hours and cumulative opioid consumption at 48h will be recorded following surgery
Quadriceps weakness | In the 48 hours following surgery
  Quadriceps weakness will be assessed at 6 and 24th hours after surgery. The patient will be asked to extend the knee with the hip flexed at 45 degrees. Quadriceps strength will be graded according to the following: Grade 0: No extension, Grade 1: Extension against gravity but not against resistance, Grade 2: Extension against gravity and resistance.
Ability to perform physiotherapy | In the 48 hours following surgery
  Ability to perform physiotherapy and whether the inability to perform physiotherapy was due to pain or motor weakness will be recorded by the physiotherapist at 24 and 48 hours after surgery

OTHER OUTCOMES:
Adverse effects | In the 48 hours following surgery
  Any occurring adverse effects due to opioid use or nerve block will be recorded should they occur.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Hospitals, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes